CLINICAL TRIAL: NCT07268027
Title: The Effect of a Constructivist-Based Prenatal Education Program on Pregnant Women's Fear of Childbirth, Pain Beliefs, and Self-Efficacy for Normal Delivery: A Randomized Controlled Trial.
Brief Title: Constructivist Prenatal Education Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Assoc. Prof. Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/1052
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Fear of Childbirth; Self-Efficacy; Childbirth Education; Pain
Keywords: Pregnancy Education Program; Fear of Childbirth; Pain Belief; Self-Efficacy for Normal Birth
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (Placebo Comparator): No additional intervention will be provided to the control group beyond the information they receive during routine prenatal care and in-service trainings, and the control group will consist of pregnant women who do not attend the prenatal school education. After the study is completed, control group participants will be offered the opportunity to attend the standard prenatal school education if they wish.
  Interventions: Other: Constructivist-Based Prenatal Education Group
- Intervention Group (Experimental): Pregnant women who agree to participate in the study and are assigned to the childbirth preparation education group will receive a Constructivist-Based Prenatal Education Program in the prenatal school department of the hospital for a total of 24 hours over 3 days. Participants in the intervention group will attend the classes in groups of 15.
  Interventions: Other: Constructivist-Based Prenatal Education Group

INTERVENTIONS:
Other: Constructivist-Based Prenatal Education Group — Pregnant women who agree to participate in the study and are assigned to the childbirth preparation education group will receive a Constructivist-Based Prenatal Education Program in the prenatal school department of the hospital for a total of 24 hours over 3 days. Participants in the intervention group will attend the classes in groups of 15.
  Other Names: Education Group

SUMMARY:
The Effect of a Constructivist-Based Prenatal Education Program on Pregnant Women's Fear of Childbirth, Pain Beliefs, and Self-Efficacy for Normal Delivery: A Randomized Controlled Trial.

DETAILED DESCRIPTION:
The study is a randomized controlled trial. It will be conducted at the prenatal school of Konya City Hospital between December 2025 and May 2026. A total of 126 primiparous pregnant women will be included in the study (intervention group n=63, control group n=63). The intervention group will receive the Constructivist-Based Prenatal Education Program, while the control group will receive the standard prenatal care and education provided by the hospital. Data will be collected using a personal information form, the Fear of Childbirth Scale, the Pain Beliefs Scale, and the Self-Efficacy for Normal Birth Scale.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the hospital's prenatal school and actively participating in the 3-day training sessions,
* Aged 18 years or older,
* Between 20 and 32 weeks of gestation,
* Having a singleton and low-risk pregnancy,
* Primiparous (expecting their first birth),
* Voluntarily agreeing to participate by signing the written informed consent form,
* Able to read, understand, and communicate in Turkish.

Exclusion Criteria:

* Those who have previously given birth vaginally or by cesarean section (multiparous women),
* Those with multiple pregnancies,
* Those who conceived through assisted reproductive techniques,
* Those diagnosed with serious obstetric or medical complications during pregnancy (such as preeclampsia, gestational diabetes, or risk of preterm birth),
* Those with a history of psychiatric diagnosis or currently receiving psychiatric treatment,
* Foreign nationals.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the sociodemographic characteristics of pregnant women before the training with a survey. | 6 months
  Sociodemographic information of pregnant women will be collected through surveys, compared, and reported.
Comparison of obstetric characteristics of pregnant women before the training with a questionnaire. | 6 months
  Obstetric data of pregnant women will be collected through questionnaires, compared, and reported.
Comparison of the means of the Fear of Childbirth Scale among pregnant women across groups. | 6 months
  The Fear of Childbirth Scale will be administered to pregnant women. The Respectful Childbirth Care scale ranges from 0 to 160 points (min-max), with higher scores indicating higher fear of childbirth.
Comparison of the Pain Beliefs Scale means among pregnant women across groups. | 6 months
  The Pain Beliefs Scale will be administered to pregnant women.The scale evaluates two types of pain-related beliefs: organic and psychological. It includes 12 items rated on a 6-point Likert scale, with 8 items assessing organic beliefs (pain as a physiological or pathophysiological condition) and 4 items assessing psychological beliefs (pain influenced by anxiety, depression, or external factors). No total score is calculated; each subscale score is the mean of its items. Higher scores indicate stronger beliefs in that specific dimension.
Comparison of mean scores on the Self-Efficacy Scale for Normal Childbirth among pregnant women across groups. | 6 months
  The Self-Efficacy Scale for Normal Childbirth will be administered to pregnant women. Possible scores on the scale are 0-90 (min-max). Higher scores indicate higher self-efficacy levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Seyhan Çankaya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No